CLINICAL TRIAL: NCT00572585
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Design Study to Explore the Efficacy, Safety and Tolerability of AEB071 in Patients With Active, Moderate to Severe Ulcerative Colitis
Brief Title: Efficacy, Safety and Tolerability of AEB071 in Patients With Active, Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAEB071A2210; 2007-002542-38
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2017-03

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; immunosuppressive therapy; AEB071; Modified Baron score; Partial Mayo score
MeSH Terms: conditions — Colitis, Ulcerative | interventions — sotrastaurin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AEB071 (Experimental)
  Interventions: Drug: AEB071
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AEB071
  Arms: AEB071
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of AEB071 in the treatment of active, moderate to severe ulcerative colitis in patients who have failed conventional therapy using mesalamine or steroids

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years males and females
* Female subjects of childbearing potential must be using two methods of contraception
* Active, moderate to severe disease
* Poor response to or no toleration of conventional therapy (e.g. steroids, mesalamine)
* Good communication with the investigator, understanding and compliance with the requirements of the study and written informed consent

Exclusion Criteria:

* Allergy to the drug
* Very low or high body weight
* Ongoing treatment with specific other medication (e.g. antibiotics)
* Diagnosis of primary sclerosing cholangitis
* Renal impairment
* Toxic megacolon
* Presence or history of specific other diseases, cancer, cardiac abnormalities, abnormal laboratory findings
* History of alcohol or drug abuse
* Pregnant or breastfeeding women
* Positive HIV, Hepatitis B or Hepatitis C test result

Other protocol-defined inclusion/exclusion criteria do apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Rate of induction of remission after 28 days of treatment (using the Partial Mayo Score and the Modified Baron Score), also an Endoscopic biopsy will be taken | Partial Mayo Score throughout entire study, biopsy at end of dosing period

SECONDARY OUTCOMES:
Safety and tolerability assessments (vital signs, electrocardiogram [ECG], blood samples, serious adverse events, adverse events) | Throughout entire study
Measurement of drug concentrations in blood | During the dosing period only
Relationship between drug concentration in blood and disease activity | Dosing period only

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- United States (7):
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Lafayette, Louisiana
  - Novartis Investigative Site, Chesterfield Twp, Michigan
  - Novartis Investigative Site, Troy, Michigan
  - Novartis Investigative Site, Oklahoma City, Oklahoma
- Denmark (2):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Odense C
- Germany (9):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Stuttgart
- Poland (2):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Poznan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CAEB071A2210 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8363